CLINICAL TRIAL: NCT00900965
Title: A Pilot Study on the Effect of Electroacupuncture on Functional Brain Mapping in Patients With Irritable Bowel Syndrome
Brief Title: Effect of Electroacupuncture in Patients With Irritable Bowel Syndrome
Acronym: IBS_FBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Prof Winnie C.W. Chu, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBS_FBM
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; IBS; fMRI; acupuncture; functional; brain
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electroacupuncture treatment (Active Comparator): A specially designed copper needle (0.22 x 4 mm), which can be used safely in MRI suite, will be inserted through a plaster over the respective acupoints, under which a plastic ring will be positioned, connected with electrical stimulation machine (EY-3308 Model, G6805-2 Mayfair) through wires with stimulation frequency of 150 Hz, lasting for 30 minutes.
  Interventions: Device: Electroacupuncture treatment (electrical stimulation machine (EY-3308 Model, G6805-2 Mayfair))
- Sham acupunture treatment (Sham Comparator): Needle will be positioned at 2 cm away from the true respective acupoints, with a blunted, telescopic placebo needle. The same electric stimulation will be the same as real acupuncture treatment.
  Interventions: Device: Sham acupuncture treatment (electrical stimulation machine (EY-3308 Model, G6805-2 Mayfair))

INTERVENTIONS:
Device: Electroacupuncture treatment (electrical stimulation machine (EY-3308 Model, G6805-2 Mayfair)) — A specially designed copper needle (0.22 x 4 mm), which can be used safely in MRI suite, will be inserted through a plaster over the respective acupoints, under which a plastic ring will be positioned, connected with electrical stimulation machine (EY-3308 Model, G6805-2 Mayfair) through wires with stimulation frequency of 150 Hz, lasting for 30 minutes.
  Other Names: electrical stimulation machine (EY-3308 Model, G6805-2 Mayfair)
  Arms: Electroacupuncture treatment
Device: Sham acupuncture treatment (electrical stimulation machine (EY-3308 Model, G6805-2 Mayfair)) — Needle will be positioned at 2 cm away from the true respective acupoints, with a blunted, telescopic placebo needle. The same electric stimulation will be the same as real acupuncture treatment.
  Arms: Sham acupunture treatment

SUMMARY:
Irritable bowel syndrome (IBS) is the most common digestive disorder that affects more than 5% of population in Hong Kong. However, there is no effective treatment of IBS using Western Medicine. Acupuncture, a traditional therapeutic modality, has been used in China for thousands of years for various pain disorders. In addition to analgesia, acupuncture has also been shown to influence physiology of gastrointestinal tract. The investigators set out to evaluate the therapeutic value of acupuncture in IBS. The investigators will study its effects on rectal sensation and brain activity in patients with IBS.

All patients will be evaluated for study eligibility at visit 1 (baseline). Baseline assessment includes individual IBS symptoms (pain/discomfort, bloating, constipation, and diarrhea) as perceived by patients will be scored. The syndrome of IBS patients will also be recorded and analyzed based on the Chinese medicine theories. All patients will then undergo baseline rectal barostat for thresholds of rectal sensation. At visit 2, eligible patients will be randomly assigned to either (1) electroacupuncture or (2) sham electroacupuncture treatment groups. Functional Magnetic Resonance Imaging (fMRI) scanning will be performed before, during and after the electroacupuncture or sham electroacupuncture treatment.

DETAILED DESCRIPTION:
All patients will be evaluated for study eligibility at visit 1 (baseline). Baseline assessment includes the following items:

1. Global symptom assessment: Based on Rome III Working Group recommendation, a clinical outcome response measure is used in which patients are required to report "improved", "the same" or "worsened" to the question "Do you have adequate symptom relief in the past 7 days?"
2. Individual IBS symptoms: The individual IBS symptom (pain/discomfort, bloating, constipation, and diarrhea) as perceived by patients will be scored in a 5-point scale (0=none or asymptomatic; 1=mild with no limitation of normal activities; 2=moderate with limitation of some normal activities; 3=intense and unable to carry out most normal activities; 4=incapacitating symptom that are intolerable and unable to carry out all normal activities).
3. Syndrome of Chinese medicine: The syndrome of IBS patients will be recorded and analyzed based on the Chinese medicine theories. These symptoms involving: fatigue, appetite, sense of mouth, quality of sleep, the coating of tongue, pulse, etc.
4. Quality of life (QOL) assessment: A disease-specific questionnaire- IBS Quality of Life Scale (Chinese) will be used for assessment of QOL in response to treatment. The questionnaire was locally validated, and was recently developed by our group.
5. Rectal barostat: The patients will be evaluated for the sensory threshold and maximum tolerable threshold of rectum in response to balloon distension of rectum before the acupuncture treatment.

At visit 2, eligible patients will be randomly assigned to either (1) electroacupuncture or (2) sham electroacupuncture. During the treatment, the patient will receive fMRI to evaluate the cerebral cortical activity in response to balloon distension of rectum. Three sets of real-time functional brain mapping using fMRI will be performed during rectal balloon distensions at maximum tolerable pressure at the following time points:

1. 10 minutes after acupuncture needle insertion before delivery of electrical stimulation
2. 15 minutes after electrical stimulation begins (electrical stimulation continues during MRI)
3. Immediately after electrical stimulation stops before removal of acupuncture needle

Rectal barostat:

The barostat device contains a built-in computer system that can be programmed to automatically perform distensions of balloon with fixed time lags and bag pressure increments. Variation in balloon volume in a constant pressure reflects the change in tone and compliance of the visceral wall. Furthermore, through a programmed variation in intraballoon pressure, the sensory threshold of subject can be evaluated.

The patient is instructed to take low residue diet 2 days prior to barostat. On the day before barostat, bowel preparation is performed by ingestion of 4 liters of polyethylene glycol solution in 2 divided doses. After a 12-hour fast, the participant is positioned in supine position on MRI table. A barostat bag is inserted into the rectum. The barostat device is connected to the barostat catheter using a low compliance PVC tubing. The participant will remain alone in MRI cubicle during the whole experiment but a speaker and microphone system allows communication with the investigator. He/she is also provided a squeeze bulb to signify pain. Repeated squeezing of the bulb signifies request for termination of procedure.

Phasic isobaric rectal distensions are performed automatically using ascending method of limits (AML) protocol with successive increments of 4 mm Hg (40-second duration) alternating with intermittent periods of bag deflation (40 seconds). During each distension phase, the participant is requested to report the perception ratings by pressing on the perception panel of barostat device with the following scale: (1) no sensation (2) the first sensation of balloon distension, (3) desire for defecation, (4) maximum tolerable sensation. The procedure will be stopped when pain or maximum tolerable sensation is reported. The sensory threshold is defined as lower limit of the bag pressure that evokes the first sensation of balloon distension. The pain threshold is defined as pressure that elicits a "pain" response or maximum tolerable sensation.

Electroacupuncture Treatment:

Treatment will be performed by a single licensed acupuncturist. Both the patient and the investigator are unaware of the treatment assigned. A specially designed copper needle (0.22x4mm), which can be used safely in MRI suite, will be inserted through a plaster over the respective acupoints, under which a plastic ring will be positioned, connected with electrical stimulation machine (EY-3308 Model, G6805-2 Mayfair) through wires with stimulation frequency of 150Hz, lasting for 30 minutes. For sham acupuncture, the needle will be positioned at 2cm away from the true respective acupoints., the same electric stimulation will be the same as real acupuncture treatment. The treatment will be given by an independent acupuncturist who is not involved in the data acquisition and analysis. Points for acupuncture treatment are chosen to regain the balance of liver qi stagnation and strengthen the spleen:

Anatomical location (Function according to TCM)

1. SP06:3cm above the medial malleolus dorsal tibial rim (Strengthens spleen and stomach)
2. ST25:2cm lateral to the umbilicus (Strengthens spleen and stop diarrhea)
3. ST36:5cm below patella, 2 cm lateral of the tibial rim (Strengthens spleen and stomach)
4. ST37:3cm below ST36 (Strengthens spleen and stop diarrhea)

Functional MRI:

BOLD imaging is performed with a 3-T MRI scanner (Philips Achieva 3.0T, X series, Quasar Dual MRI system). Each study consists of axial T1-weighted spin echo images (matrix of at least 192 × 256) covering the whole brain for anatomical correlation. Functional scan is performed using a single-shot echo planar pulse sequence in an interleaved multislice format with a field of view of 24 cm and a matrix size of at least 64 × 64, resulting in a in-plane resolution of 3.75 × 3.75. The pulse sequence parameters include a 90° flip-angle with a TE (time to echo)/TR (repetition time) of 60 ms/4000 ms. Each paradigm consists of 5 periods. Each period will consist of rest and stimulation (tube inflation causing rectal distension). In each period, 50 dynamics are performed. Each dynamic will last for 2 seconds. The scans will be performed with the rectal tube inflated to render:

1. Desire for defecation, and
2. Painful sensation, as determined by the barostat study at baseline visit within one week before MRI scanning.

ELIGIBILITY:
Inclusion Criteria:

* Irritable bowel syndrome of diarrhea type as defined by Rome III criteria
* Age 18-65 years
* Normal colonic evaluation within 12 months (with either colonoscopy or barium study)

Exclusion Criteria:

* IBS-constipation, mixed or unsubtyped
* Pregnancy
* Medical history of organic colonic bowel disease
* History of sensitivity to acupuncture
* Psychiatric or additive disorder
* Patients who have received acupuncture in the past 6 months
* Concomitant medications including anti-diarrhea agent, anti-depressant, narcotic analgesic and anti-cholinergic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Sensory and pain thresholds as determined by rectal barostat | At baseline study visit
Degree of cortical activation as determined by functional MRI | At study visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Winnie C.W. Chu, MBChB, FRCR, MD, FHKAM, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin, Hong Kong, China